CLINICAL TRIAL: NCT03315754
Title: Study of the Efficacy, Safety and Quality of Life After TOOKAD® Soluble Vascular Targeted Photodynamic Therapy (VTP) for Minimally Invasive Treatment of Localized Intermediate Risk Prostate Cancer.
Brief Title: Study of the Efficacy, Safety and Quality of Life After TOOKAD® Soluble (VTP) for Intermediate Risk Prostate Cancer.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN1601 PCM204
Record Dates: First submitted 2017-10-02; First posted 2017-10-20 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-10

CONDITIONS: Localized Prostate Cancer
MeSH Terms: interventions — padeliporfin

STUDY DESIGN:
Intervention Model Description: Single center, single-arm, open-label, 60-month follow-up phase IIb clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TOOKAD Soluble 4 mg/kg (Experimental): TOOKAD® Soluble VTP treatment consist of the combination of a single, 10-minute IV infusion of TOOKAD® Soluble at the dose of 4 mg/kg, followed by the illumination of the zone to be treated with a 753-nm laser light delivered through transperineal interstitial optical fibers at a power of 150 mW/cm and light energy of 200 J/cm applied over 22 minutes and 15 seconds.
  Interventions: Drug: TOOKAD Soluble 4 mg/kg

INTERVENTIONS:
Drug: TOOKAD Soluble 4 mg/kg — Vascular targeted photodynamic therapy using TOOKAD Soluble
  Other Names: WST11

SUMMARY:
Single center, single-arm, open-label, 60-month follow-up phase IIb clinical trial. Men with localized prostate cancer will receive TOOKAD® Soluble VTP under general anesthesia.

To evaluate the absence of biopsy detectable Gleason grade 4 or 5 prostate cancer tumors anywhere in the prostate gland on 12-month, post-treatment biopsy following TOOKAD® Soluble-VTP in men with prostate cancer Gleason score 7(3+4).

DETAILED DESCRIPTION:
This is a single center, single-arm, open-label, 60-month follow-up phase IIb clinical trial. The primary objective of the study is to evaluate the absence of biopsy detectable Gleason grade 4 or 5 prostate cancer tumors anywhere in the prostate gland on 12-month, post-treatment biopsy following TOOKAD® Soluble-VTP. Men with Gleason score 7 (3+4) prostate cancer on one half of the prostate will receive TOOKAD® Soluble VTP under general anesthesia. Treatment will consist in hemiablation procedure designed to destroy the lobe of the prostate gland that contains the Gleason score 7 (3+4) cancer. Afterwards, patients will be followed for 5 years (60 months) with clinical evaluation, questionnaires on QOL, erectile and urinary functions, and PSA testing. In addition, treatment outcomes will be assessed based on prostate biopsy results at 3, 12, 24, 36, 48 and 60 months after the TOOKAD® Soluble treatment. All patients will undergo biopsy at 3 and 12 months. If the Month 3 biopsy is positive for any cancer, patients will be allowed a single re-treatment by TOOKAD® Soluble VTP to one or both lobes.

ELIGIBILITY:
Inclusion Criteria:

1. Men over 18 years of age.
2. Patients who have had a multiparametric MRI of the prostate performed and have undergone transrectal systematic biopsy plus biopsy of any volumes considered suspicious per the MRI (PIRADS version 2 score of 4 or 5) within 6 months before signing consent.
3. Histologic diagnosis of prostate cancer identifying Gleason score of 3+4 on one half of the prostate gland in no more than 2 sextants of the prostate gland and not present in more than 50% of any one core taken systematically. The involvement criterion does not apply to cores taken from MRI suspicious volumes.
4. Patients with concomitant Gleason score 3+3 prostate cancer in less than 50% of any core at any site will be considered eligible.
5. Prostate cancer stage up to cT2a - N0/Nx - M0/Mx.
6. Prostate volume ≥25 mL and ≤70 mL.
7. Serum PSA ≤10 ng/mL.
8. Men who are sexually active with women of childbearing potential must use contraceptive method with a failure rate of less than 1% per year. Contraception should be continued for a period of 90 days after the VTP procedure. The individual methods of contraception may be determined in consultation
9. Signed Informed Consent Form.

Exclusion Criteria:

1. Unwillingness to accept the treatment;
2. Any prior or current treatment for prostate cancer, including surgery, radiation therapy (external or brachytherapy) or chemotherapy;
3. Any surgical intervention for benign prostatic hypertrophy;
4. Any condition or history of illness or surgery that might pose an additional risk to men undergoing the VTP procedure;
5. Life expectancy less than 10 years;
6. Participation in another clinical study involving an investigational product within 1 month before study entry;
7. Inability to understand the informed consent document, to give consent voluntarily or to complete the study tasks, especially inability to understand and fulfill the health-related QOL questionnaire;
8. Subjects in custody and or residing in a nursing home or rehabilitation facility;
9. Biopsy proven locally advanced or metastatic prostate cancer.
10. Any condition or history of illness or surgery that in the opinion of the investigator might affect the conduct and results of the study or pose additional risks to the subject (e.g., cardiac or respiratory disease precluding general anesthesia; anticoagulant treatment which cannot be temporarily withdrawn for the procedure).
11. Medical conditions that preclude the use of general anesthesia;
12. Any condition or history of active rectal inflammatory bowel disease or other factors which might increase the risk of fistula formation;
13. Hormonal manipulation (excluding 5-alpha-reductase inhibitors) that alters androgen production within the previous 6 months;
14. History of urethral stricture disease;
15. History of acute urinary retention within 6 months of study entry;
16. Condition requiring medication with potential photosensitizing effects (tetracyclines, quinolones, sulphonamides, phenothiazines, sulfonylurea hypoglycaemic agents, thiazide diuretics, griseofulvin, and amiodarone) if these treatments could not be stopped at least 10 days before and for 3 days after the VTP procedure or replaced by treatments without photosensitizing properties;
17. Anticoagulant drugs (e.g., warfarin) that could not be withdrawn during the 10 days prior to the VTP procedure or antiplatelet drugs (e.g. aspirin) that could not be withdrawn during the 10 days prior to the VTP procedure and 3 days after VTP;
18. Renal and hepatic disorders with values of >1.5 times the upper limit of normal (ULN) or blood disorders (upon clinician judgment);
19. A history of sun hypersensitivity or photosensitive dermatitis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2025-02-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty men presenting with Gleason score 7 (3+4) prostate cancer in at least one lobe were enrolled in the study.
Period: Overall Study
Arm/Group | TOOKAD Soluble 4 mg/kg
Started | 50
Completed | 48
Not Completed | 2
Not completed — COVID-19 complications leading to death | 1
Not completed — insurance coverage issue | 1

BASELINE CHARACTERISTICS:
Arm/Group | TOOKAD Soluble 4 mg/kg
Number analyzed (Participants) | 50
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 61.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, (%): Unknown/Not Reported | 8
  Race, (%): White | 39
  Race, (%): African American | 1
  Race, (%): Asian | 1
  Race, (%): American Indian/Alaska Native | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Number of Participants with Biopsy for Gleason score 7 (3+4) prostate cancer in at least one lobe [Count of Participants; unit: Participants] | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Biopsy for Gleason Grade 4 or 5 Prostate Cancer on 12-month Post-treatment
Description: Binary response to treatment defined as absence of Gleason grade 4 or 5 on biopsy on 12-month post-treatment following TOOKAD® Soluble VTP in men with Gleason score 7 (3+4) prostate cancer
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | TOOKAD Soluble 4 mg/kg
Number analyzed (Participants) | 45
participants | 38

2. Secondary Outcome: Absence of Gleason Grade 4 or 5
Description: Binary response to treatment defined as the absence of any Gleason grade 4 or 5 biopsy on or before months 24, 36, 48 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of gleason grade 4 or 5, the subject will be considered to have responded;
Time Frame: months 24, 36, 48 and 60
Reporting Status: Not Posted

3. Secondary Outcome: Absence of Any Prostate Cancer on Biopsy
Description: Binary response to treatment defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36 and 60. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded;
Time Frame: months 3, 12, 24, 36 and 60
Reporting Status: Not Posted

4. Secondary Outcome: Absence of Any Gleason 4 or 5 in the Treated Lobe
Description: Binary response to treatment defined as the absence of any Gleason grade 4 or 5 biopsy on or before months 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of gleason grade 4 or 5, the subject will be considered to have responded;
Time Frame: months 12, 24, 36, 48 and 60
Reporting Status: Not Posted

5. Secondary Outcome: Absence of Any Prostate Cancer on Biopsy in the Treated Lobe
Description: Binary response to treatment defined as the absence of any prostate cancer on biopsy on or before months 3, 12, 24, 36, 48 and 60 in the treated lobe. If a subject is retreated following a positive biopsy at 3 months and subsequent biopsy shows absence of any cancer, the subject will be considered to have responded
Time Frame: months 3, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

6. Secondary Outcome: Changes in Biopsy Parameters (Gleason Score)
Description: Changes in biopsy parameters (Gleason score) between the baseline biopsy and Month 3, Month12, Month 24, Month 36, Month48 and Month 60 biopsies
Time Frame: months 3, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

7. Secondary Outcome: Changes in Biopsy Parameters (Number of Positive Score)
Description: Changes in biopsy parameters (number of positive score) between the baseline biopsy and Month 3, Month12, Month 24, Month 36, Month48 and Month 60 biopsies
Time Frame: months 3, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Biopsy Parameters (Cancer Core Length)
Description: Changes in biopsy parameters (cancer core length) between the baseline biopsy and Month 3, Month12, Month 24, Month 36, Month48 and Month 60 biopsies
Time Frame: months 3, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

9. Secondary Outcome: IPSS Questionnaire
Description: Changes in patients' reported outcome measures (PROMs) for urinary symptoms using IPSS (changes in IPSS scores from baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months after treatment)
Time Frame: months 1, 3, 6, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

10. Secondary Outcome: IIEF15 Questionnaire
Description: Changes in patients' reported outcome measures (PROMs) for erectile function using IIEF 15 (changes in IIEF 15 scores from baseline to 1, 3, 6, 12, 24, 36, 48 and 60 months after treatment)
Time Frame: months 1, 3, 6, 12, 24, 36, 48 and 60
Reporting Status: Not Posted

11. Secondary Outcome: Severe Prostate Cancer-related Events
Description: Severe prostate cancer-related events: cancer extension to T3, metastasis or prostate cancer-related death
Time Frame: Up to 60 months
Reporting Status: Not Posted

12. Secondary Outcome: Secondary Prostate Cancer Treatment
Description: Use of secondary prostate cancer treatment following VTP will include surgical removal of the prostate gland, radiation treatment to the prostate gland, use of hormone or chemotherapies
Time Frame: Up to 60 months
Reporting Status: Not Posted

13. Secondary Outcome: Adverse Events
Description: Collection Adverse events
Time Frame: Up to 60 months
Reporting Status: Not Posted

14. Secondary Outcome: PSA
Description: Serum PSA measurements in ng/mL.
Time Frame: Months 1, 3, 6, 12, 24, 36, 48, 60
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: All patients experienced at least one AE during the first 12 months period of this study. A total of 379 AEs were reported, none which were related to the study drug.
Arm/Group | TOOKAD Soluble 4 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 9/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | TOOKAD Soluble 4 mg/kg (N=50)
COVID-19 (Infections and infestations) | 1/9 (1) — Patient contracted the SARS-CoV-19 and subsequently passed on after suffering Grade V symptoms. Patient data were excluded from the analyses, as the patient expired before undergoing the Month 12 evaluation.
Total knee replacement (Surgical and medical procedures) | 2/9 (2) — Grade I and III, unrelated to treatment or to the procedure
Nausea (Gastrointestinal disorders) | 1/9 (1) — Grade I
Dizziness (Nervous system disorders) | 1/9 (1) — Grade 1
Vomiting (Gastrointestinal disorders) | 1/9 (1) — Grade I
Chills (General disorders) | 1/9 (1) — Grade I
Flank pain (Musculoskeletal and connective tissue disorders) | 1/9 (1) — Grade I
Constipation (Gastrointestinal disorders) | 1/9 (1) — Grade II
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TOOKAD Soluble 4 mg/kg (N=50)
Micturition urgency (Renal and urinary disorders) | 38 (42)
Pollakiuria (Renal and urinary disorders) | 37 (41)
Hematuria (Renal and urinary disorders) | 33 (37)
Urinary tract pain (Renal and urinary disorders) | 31 (33)
Urinary incontinence (Renal and urinary disorders) | 9 (9)
Urinary tract obstruction (Renal and urinary disorders) | 7 (7)
Urinary retention (Renal and urinary disorders) | 4 (4)
Erectile dysfunction (Reproductive system and breast disorders) | 23 (25)
Haematospermia (Reproductive system and breast disorders) | 15 (17)
Perineal pain (Reproductive system and breast disorders) | 8 (8)
Edema genital (Reproductive system and breast disorders) | 4 (4)
Retrograde ejaculation (Reproductive system and breast disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 22 (24)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Proctalgia (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 16 (19)
Fatigue (General disorders) | 10 (10)
Pyrexia (General disorders) | 5 (6)
Chills (General disorders) | 3 (4)
Infections and infestations (Infections and infestations) | 11 (13)
Epididymitis (Reproductive system and breast disorders) | 3 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 (13)
Contusion (Injury, poisoning and procedural complications) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03315754/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT03315754/SAP_001.pdf